CLINICAL TRIAL: NCT01373034
Title: The Effects of Soy Dietary Fiber in Adults With Diarrhea Predominant Irritable Bowel Syndrome: Double-blind, Randomized, Placebo-controlled, Cross Over Clinical Trial
Brief Title: The Effects of Soy Dietary Fiber in Adults With Diarrhea Predominant Irritable Bowel Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Kyoung Sup Hong, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHUNG_SOY
Record Dates: First submitted 2011-06-13; First posted 2011-06-14 (Estimated); Last update posted 2011-06-14 (Estimated); Status verified 2011-06

CONDITIONS: Diarrhea Predominant Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Soy Dietary Fiber (Experimental)
  Interventions: Dietary Supplement: Soy Dietary Fiber
- Rice powder (Placebo Comparator)
  Interventions: Dietary Supplement: Rice powder

INTERVENTIONS:
Dietary Supplement: Soy Dietary Fiber — Soy Dietary Fiber, Once a day, before meal, 1 pack(20g), per oral with water 90mL
  Arms: Soy Dietary Fiber
Dietary Supplement: Rice powder — Rice powder, Once a day, before meal, 1 pack(20g), per oral with water 90mL
  Arms: Rice powder

SUMMARY:
The investigators will evaluate the efficacy of soy dietary fiber in adults with diarrhea predominant irritable bowel syndrome.

ELIGIBILITY:
Inclusion Criteria:

* willing to consent/undergo necessary procedures
* between the age of 19 and 75 years
* diarrhea predominant irritable bowel syndrome (satisfied with Rome II criteria)

Exclusion Criteria:

* uncontrolled hypertension (Blood pressure > 170/100 mmHg)
* uncontrolled diabetes mellitus (FBS > 180 mg/dL)
* malignancy, cerebrovascular disease, cardiovascular disease
* history of abdominal surgery except appendectomy and hernia repair
* inflammatory bowel disease
* clinically or laboratory-confirmed gastroenteritis
* the use of motility drug or dietary fiber supplement in 2 weeks
* allergy to soy fiber
* serum Cr > 2 x Upper normal limit
* AST or ALT > 2 x Upper normal limit
* Pregnancy, Lactating woman

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
sum of irritable bowel syndrome symptom score | after 4 weeks
  abdominal pain / abdominal discomfort urgency tenesmus abdominal distension

SECONDARY OUTCOMES:
irritable bowel syndrome symptom score | after 2 weeks and 4 weeks
  abdominal pain / abdominal discomfort urgency tenesmus abdominal distension
Stool frequency and form | after 2 weeks and 4 weeks
  Stool frequency (greater than 3 bowel movements/day or less than 3 bowel movements/week) Stool form (lumpy / hard or loose / watery stool)
Symptom control of irritable bowel syndrome | after 2 weeks and 4 weeks
Improvement of overall symptom in patient with irritable bowel syndrome | after 2 weeks and 4 weeks
Severity of overall symptom in patient with irritable bowel syndrome | after 2 weeks and 4 weeks
Severity of diarrhea | after 2 weeks and 4 weeks
Assessment for quality of life related with irritable bowel syndrome | after 2 weeks and 4 weeks
Assessment for patient satisfaction after administration completion | after 2 weeks and 4 weeks
  Overall satisfaction for treatment Whether the patient will keep up treatment

CONTACTS AND LOCATIONS:
Overall Officials: Joo Sung Kim, M.D., PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea